CLINICAL TRIAL: NCT06945367
Title: Impact of Active Learning on Beliefs, Attitudes, Perceived Skills, and Application of Evidence-Based Practice in Undergraduate Physiotherapy Students
Brief Title: Active Learning and EBP Competency in Undergraduate Physiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de la Matanza (Other)
Responsible Party: Principal Investigator, Mauro Federico Andreu, PhD, Universidad Nacional de la Matanza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UNLaM-AL
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Health Education
Keywords: Evidence-Based Practice; Health Knowledge, Attitudes, Practice; Physical Therapy Specialty; Education, Professional
MeSH Terms: conditions — Health Education; Behavior

STUDY DESIGN:
Intervention Model Description: Pre-post quasi-experimental design without a control group
Masking Description: Due to the nature of the study, blinding was not feasible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Learning Group (Experimental): Participants in this arm are fourth-year undergraduate physiotherapy students enrolled in a Research Methods course. They will receive a four-month educational intervention based on active learning strategies, including weekly group-based activities such as literature search, critical appraisal, structured presentations, peer feedback, and formative assessment using rubrics. The aim was to improve beliefs, attitudes, perceived skills, and frequency of use of evidence-based practice.
  Interventions: Behavioral: Active Learning-Based Research Methods Course

INTERVENTIONS:
Behavioral: Active Learning-Based Research Methods Course — A four-month educational intervention based on active learning strategies, delivered as part of a Research Methods course for fourth-year undergraduate students in physiotherapy. The intervention included weekly group activities focused on literature retrieval, critical appraisal, oral presentations, peer feedback, and structured formative assessments using rubrics. The aim was to improve beliefs, attitudes, perceived skills, and frequency of use of evidence-based practice.
  Other Names: AL-EBP

SUMMARY:
This study aims to evaluate the effect of an active learning-based educational intervention on competencies related to evidence-based practice (EBP) in undergraduate physiotherapy students. The intervention was embedded within a four-month Research Methods course and focused on small group activities involving literature search, critical appraisal, oral presentations, and formative assessment through rubrics.

The study follows a pre-post quasi-experimental design without a control group. Primary outcomes include students' beliefs, attitudes, perceived skills, and frequency of EBP application, assessed through a custom-developed and validated questionnaire. Secondary outcomes include academic engagement, measured using the Utrecht Work Engagement Scale - Student Version (UWES-S), and student satisfaction with the educational approach, measured using the Student Outcomes Survey. Data were collected at baseline, post-intervention, and one week after course completion.

DETAILED DESCRIPTION:
This quasi-experimental study without a control group will be conducted at the Universidad Nacional de La Matanza (UNLaM), Argentina, between March and July 2025. The study aimed to evaluate the effect of an educational intervention based on active learning strategies on evidence-based practice (EBP) competencies among physiotherapy students.

The intervention was implemented as part of a four-month Research Methods course and included weekly group-based activities such as literature retrieval, critical appraisal, oral presentations, peer feedback, and structured assessments using rubrics. The course aimed to strengthen students' beliefs, attitudes, perceived skills, and frequency of use related to EBP.

Outcomes were assessed using a custom-developed and validated questionnaire covering four domains and key competencies in EBP. Secondary outcomes included academic engagement, measured with the Utrecht Work Engagement Scale - Student Version (UWES-S), and student satisfaction, assessed through the Student Outcomes Survey. Data collection occurred at baseline, at the end of the course, and one week after completion. The study followed TREND reporting guidelines and was approved by the institutional research ethics committee at UNLaM.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students enrolled in the Research Methods course at the Universidad Nacional de La Matanza during the March-July 2024 term.
* Provided written informed consent.
* Attended at least 80% of course sessions.

Exclusion Criteria:

* Students who withdrew from the course before completion of the follow-up period.
* Incomplete or missing baseline or final evaluation data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Beliefs about Evidence-Based Practice | Baseline and immediately after the 4-month intervention
  Assessed as part of a custom-developed and validated questionnaire covering four domains and EBP-related competencies. Items were rated on a 5-point Likert scale.
Attitudes toward Evidence-Based Practice | Baseline and immediately after the 4-month intervention.
  Assessed as part of a custom-developed and validated questionnaire covering four domains and seven EBP-related competencies. Items were rated on a 5-point Likert scale
Perceived Evidence-Based Practice Skills | Baseline and immediately after the 4-month intervention.
  Assessed as part of a custom-developed and validated questionnaire covering four domains and EBP-related competencies. Items were rated on a 5-point Likert scale.
Frequency of Evidence-Based Practice Application | Baseline and immediately after the 4-month intervention.
  Assessed as part of a custom-developed and validated questionnaire covering four domains and seven EBP-related competencies. Items were rated on a 5-point Likert scale

SECONDARY OUTCOMES:
Academic Engagement | Baseline and immediately after the 4-month intervention.
  Measured using the Utrecht Work Engagement Scale - Student Version (UWES-S), a validated 9-item instrument assessing three dimensions: vigor, dedication, and absorption. Each item is rated on a 7-point Likert scale ranging from 0 ("never") to 6 ("always")
Student Satisfaction with Teaching and Assessment | One week after the completion of the 4-month intervention.
  Measured using the Student Outcomes Survey (Fieger, 2012), which includes 20 closed-ended items rated on a 5-point Likert scale. The scale is organized into three domains: satisfaction with teaching (items 1-6), assessment methods (items 7-11), and learning experience (items 12-19). Item 20 assesses overall satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional de la Matanza, San Justo, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No